CLINICAL TRIAL: NCT00986505
Title: Effect of Intravenous Lidocaine on Manifestations of Fibromyalgia
Brief Title: Intravenous Lidocaine for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Roberto Vlainich, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IV lidocaine
Record Dates: First submitted 2009-08-03; First posted 2009-09-30 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Fibromyalgia
Keywords: lidocaine; fibromyalgia; intravenous lidocaine; manifestations
MeSH Terms: conditions — Fibromyalgia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lidocaine (Experimental): Comparison between intravenous lidocaine and saline infusion
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Intravenous lidocaine once a week
  Other Names: Lidocaine infusion; Saline infusion

SUMMARY:
The effect of intravenous lidocaine infusion on manifestations of fibromyalgia manifestations were recorded before and 4 weeks after treatment. Pain intensity was rated on a numerical scale.The combination of 240 mg intravenous lidocaine (once a week) and 25 mg amitriptyline for 4 weeks did not modify pain intensity or manifestations in patients with fibromyalgia.

DETAILED DESCRIPTION:
Thirty patients ranging in age from 18 to 60 years, with fibromyalgia (American College of Rheumatology criteria: pain in the four quadrants of the body for at least 3 months and a minimum of 11 out of 18 tender points) were studied. Other manifestations were also recorded: sleep disorders, fatigue, subjective edema, depression, and paresthesia.

Criteria for exclusion were alterations in thyroid, rheumatological, renal and hepatic function; trauma; rheumatic, neuromuscular or psychiatric disease; infectious arthropathy; other pain syndromes; drug hypersensitivity, and pregnancy.

All patients received amitriptyline at a dose of 12.5 mg in the first week and 25 mg over the subsequent 4 weeks. Patients of group 1 (n = 15) received 125 mL 0.9% saline and patients of group 2 (n = 15) received 240 mg lidocaine diluted in 125 mL 0.9% saline. The solutions were infused over a period of 1 h, once a week, for 4 weeks (T1, T2, T3 and T4).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years, with fibromyalgia (American College of Rheumatology criteria: pain in the four quadrants of the body for at least 3 months and a minimum of 11 out of 18 tender points

Exclusion Criteria:

* Thyroid, rheumatological, renal and hepatic function
* Trauma
* Rheumatic, neuromuscular or psychiatric disease
* Infectious arthropathy
* Other pain syndromes
* Drug hypersensitivity; AND
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
pain | 1day

SECONDARY OUTCOMES:
other signs | 1day

CONTACTS AND LOCATIONS:
Overall Officials: Rioko K Sakata, MD, PhD, Study Director — Universidade Federal de São Paulo